CLINICAL TRIAL: NCT06314165
Title: Evaluation of the Effect of Music Medicine Application on Menstrual Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sevgi Özkan, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PamukkaleU-SBE-RND-01
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Menstruation; Syndrome
Keywords: music medicine; menstruation symptom; menstrual pain
MeSH Terms: conditions — Menstruation Disturbances; Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Two groups: comparative experiment and control
Who Masked: Participant
Masking Description: Participants included in the study will not know which group they are in. In this way, the study will be carried out in a single-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group practicing music medicine (Experimental): There will be 2 follow-ups for each group. In the first follow-up for the experimental group, when symptoms begin on the first day of their menstrual period, they will be asked to fill out the Menstruation Symptom Scale and Visual Analogue Scale, and the designated music will be played for 30 minutes. After 30 minutes, he/she will be asked to fill out the same surveys again. In the 2nd follow-up (during the menstrual period one month after the first follow-up), they will be asked to repeat what was done in the 1st follow-up on the first day of their menstrual period.
  Interventions: Other: music medicine practice
- Group where music medicine is not applied (No Intervention): Two follow-ups will be applied to the groups. At the first follow-up for the control group, they will be asked to fill out the Menstruation Symptom Scale and Visual Analog Scale when symptoms begin on the first day of their menstrual period. In the 2nd follow-up (during the menstrual period one month after the first follow-up), they will be asked to repeat what was done in the 1st follow-up on the first day of their menstrual period.

INTERVENTIONS:
Other: music medicine practice — Music medicine will be applied
  Arms: group practicing music medicine

SUMMARY:
In this study, the "Music Medicine Application" method was chosen in line with the literature and guidelines and it is aimed to determine whether it is effective in reducing the symptoms experienced by female students with "Music Medicine Application" during the menstrual period.

DETAILED DESCRIPTION:
This study aims to determine whether the application of music medicine is effective in reducing the symptoms experienced by female students during the menstrual period. The type of research was planned as a prospective, randomized controlled experimental study with a pretest-posttest control group. The research will be conducted with female students studying at Pamukkale University Faculty of Health Sciences. The data of the research will be collected between March 2024 and February 2025. Personal Information Form, Visual Analogue Scale and Menstruation Symptom Scale will be used to collect data. It was determined that a total of 62 people should participate in the research, 31 in the experimental group and 31 in the control group. As the randomization method, "simple randomization" will be used to ensure an equal number of samples in the experimental and control groups. Randomization will be done using the www.randomizer.org application. The data will be analyzed using the SPSS (23.0) package program. Continuous variables will be given as mean ± standard deviation and categorical variables will be given as number and percentage. Significance Test of Difference Between Two Means in comparing independent group differences when parametric test assumptions are met; When parametric test assumptions are not met, Mann-Whitney U test will be used to compare independent group differences.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the research
2. Menstrual cycle length has been within normal limits (21-35) for the last 3 months
3. Not using oral contraceptives for the last 3 months
4. Not having any psychiatric problems and not receiving any treatment for this in the last 3 months.
5. Not using painkillers or any pharmacological agents or methods that reduce symptoms during the study.
6. Participants who marked 1.1-10 according to Visüel analog scala

Exclusion Criteria:

1. Presence of chronic diseases or serious medical conditions
2. Presence of another physical or psychological disorder that may affect menstrual symptoms
3. Presence of psychiatric or psychological disorders
4. Active drug use or hormone therapy
5. Having given birth
6. Answering survey questions incompletely or not answering them
7. Participants who marked 0-1 according to Visüel analog scala
8. Not applying music medicine for the experimental group

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study will be conducted with female students experiencing menstruation symptoms.
Enrollment: 62 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
menstruation symptom scale | Two months
  Participants are asked to rate the symptoms they experience regarding menstruation between 1 (never) and 5 (always). Scale items are numbered according to certain factors for ease of use. Items 1-13 belong to the "Negative effects/somatic complaints" subcategory, items 14-19 belong to the "Menstrual pain symptoms" subcategory, and items 20-22 belong to the "Coping methods" subcategory. A five-point Likert type was used in the Menstruation Symptom Scale, which consists of 22 items. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the relevant sub-dimension. An increase in the mean score for sub-dimensions indicates that the severity of menstrual symptoms in that sub-dimension has increased.

SECONDARY OUTCOMES:
Visual Analogue Scale | Two months
  Participants were included in the "healthy" category when they marked the 0-1 range of the scale, and were included in the "Menstruation pain" category when they marked the 1.1-10 range. They were divided into 3 groups according to pain severity. 1.1-3: Mild pain, 3.1-7: Moderate pain, 7.1-10: Severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Özkan Professor Doctor, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University Faculty of Health Sciences, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No